CLINICAL TRIAL: NCT01344811
Title: A Randomized, Open, Parallel, Multi-center Trial to Evaluate Weight Loss Efficacy of Smart Care Service in Obese Patients With Metabolic Syndrome.
Brief Title: Effects of Telemonitoring Service for Obesity Care
Acronym: Smart-OB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Hee, Lee (Industry)
Collaborators: LG Electronics Inc. (Industry); Purdue University (Other)
Responsible Party: Sponsor-Investigator, Chang Hee, Lee, Chief Research Engineer, LG Electronics Inc.
Organization: LG Electronics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SmartCare-OB
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: telemonitoring; usual care; telehealth; home care; Health Care Quality; Access; Evaluation
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemonitoring group (Experimental): * A Smartphone, body composition analyzer and Pedometer will be provided
  * transmitting the results to the Smart Care Server via Smartphone
  * At Smart care Center,care manager will provide remote body weight and activity monitoring and individual obesity case management
  Interventions: Procedure: Telemonitoring
- Control group (Other): * A weighing scale and Pedometer will be provided
  * recording in a self diary of body weight and the number of steps
  Interventions: Other: control group

INTERVENTIONS:
Procedure: Telemonitoring — The Telemonitoring group will be provided the Smartphone, body composition analyzer and pedometer. They should visit the site once per every 3 months (12 weeks), and measure their body composition during study period. After measurement of body composition, the subjects should make transmit measured information through Smartphone into a centralized server of Smart Care Center. At Smart care Center, care manager will provide remote body composition and activity monitoring and individual obesity case management
  Other Names: Smartcare System : Telemonitoring
  Arms: Telemonitoring group
Other: control group — The control group will receive a weighting scale and pedometer. They should perform the same weight measurement (minimum three times a week) like the intervention group during the study, and measured results should be recorded in a diary of self body weight and the number of steps. In addition, the subjects should visit the site once per every three months (12 weeks).
  Other Names: Self Body Weight measurement
  Arms: Control group

SUMMARY:
A randomized, open, parallel, multi-center trial to evaluate weight loss efficacy of Smart Care Service in obese patients with metabolic syndrome.

DETAILED DESCRIPTION:
1. Objectives : To evaluate superiority of U(Ubiquitous)-Healthcare(hereinafter referred to as Smart Care) Service being combined conventional treatment with health care service, in comparison to conventional treatment in obese patients with metabolic syndrome.
2. Test and control group

   * Test groups : The subject group who is receiving health care services using conventional treatment (hospital visit) and Smart Care Service (Telemonitoring).
   * Control group : The subject group who is receiving conventional treatment (hospital visit).
3. Target Subject: Obese patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age: More than 20 years of age and under 70 years of age.
2. BMI ≥ 25kg/m2
3. Patients with metabolic syndrome (who have more than three of following 5 components of metabolic syndrome) and who are able to receive outpatient treatment.

   A. Abdominal obesity: Waist circumference≥90cm(Male), 85cm(Female) B. Patients whose blood pressure ≥130/85mmHg(systolic blood pressure over 130 or, diastolic blood pressure over 85) or patients who are taking blood pressure medication.

   C. Fasting Blood Glucose (FPG)≥ 100mg/dl. D. Patients whose triglyceride ≥150 mg/dl or patients who are taking fibrate. E. High-density lipoprotein cholesterol (HDL) < 40 mg/dl (Male), 50 mg/dl(Female)
4. Patients who are able to understand the purpose of this trial and to read and write.
5. Patients who are able to use U-healthcare Smartphone for this trial.
6. Patients who participate voluntarily and sign the informed consent.

Exclusion Criteria:

1. Type I diabetes mellitus patients and type II diabetes mellitus patients requiring insulin therapy.
2. Patients currently being hospitalized or planning to hospitalize during the study period.
3. Patients were diagnosed with myocardial infarction or stroke within 1 year
4. End Stage Renal Disease patients requiring renal replacement therapy, Serum creatinine level is greater than 1.5 times the upper limit of normal.
5. Females who are pregnant
6. Hepatic failure (severe hepatic dysfunction). Liver Function Test (AST or ALT) is greater than 3 times the upper limit of normal.
7. Uncontrolled chronic lung disease.
8. Patients with known gallstone.
9. Patients who have cognitive disorder or psychiatric problems.
10. Patients who are taking anti-obesity medications such as Reductil, Xenical, etc., or patients are planning to receive the medications.
11. Patients who are taking Synthroid, diabetes medications or psychiatric medications which may affect on body weight.
12. Any clinically significant medical condition including neurologic disease, gastrointestinal disease or malignant tumor, etc., which may affect the test results, or any other medical condition which in the opinion of the investigator makes the patients unsuitable for participation in the trial.
13. Patients who have participated in other clinical trial (except for the observational study) within 12 weeks prior to screening visit.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Weight Change from Baseline to 24 weeks | 0 and 24 weeks

SECONDARY OUTCOMES:
Body Mass Index (BMI) changes | 0 and 24 weeks
  Reduces of body mass index
  - BMI=Body weight (kg)/Height2(m)
Proportion of subjects whose body weight decreased more than 10% | 0 and 24 weeks
Changes in body fat rate | 0 and 24 weeks
  Reduces in body fat rate
Changes in waist circumference | 0 and 24 weeks
  Reduces waist circumference
Changes in lipid profile | 0 and 24 weeks
  Changes in lipid profile(total cholesterol, HDL cholesterol, LDL cholesterol triglycerides)
Changes in blood pressure | 0 and 24 weeks
  Blood pressure value when hospital visiting
  * Clinic blood pressure
  * Changes in mean Blood Pressure from baseline to 24 weeks visit
Changes in prevalence rate of metabolic syndrome | 0 and 24 weeks
Changes in the number of metabolic syndrome components | 0 and 24 weeks
  Reduce the number of metabolic syndrome components
Changes in lifestyle | 0 and 24 weeks
  Changes in lifestyle such as smoking, drinking, dietary and physical activity, etc
Patients' satisfaction | 24 weeks
  applicable to Only Telemonitoring group

CONTACTS AND LOCATIONS:
Overall Officials: Bi-Ryong Cho, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Seoul

REFERENCES:
- [Derived] Oh B, Yi GH, Han MK, Kim JS, Lee CH, Cho B, Kang HC. Importance of Active Participation in Obesity Management Through Mobile Health Care Programs: Substudy of a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Jan 3;6(1):e2. doi: 10.2196/mhealth.8719. PMID 29298749
- [Derived] Oh B, Cho B, Han MK, Choi H, Lee MN, Kang HC, Lee CH, Yun H, Kim Y. The Effectiveness of Mobile Phone-Based Care for Weight Control in Metabolic Syndrome Patients: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2015 Aug 20;3(3):e83. doi: 10.2196/mhealth.4222. PMID 26293568